CLINICAL TRIAL: NCT04608539
Title: The Postoperative Iron in Cardiac Surgery (PICS-) Trial: A Randomised Clinical Trial Comparing the Efficacy of Single-, High-dose Intravenous Iron and Oral Iron for the Treatment of Anaemia Following Cardiac Surgery
Brief Title: A Clinical Trial Assessing the Efficacy of Intravenous Iron for the Treatment of Anemia Following Cardiac Surgery
Acronym: PICS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michael Kremke (Other)
Collaborators: Aarhus University Hospital (Other); University of Aarhus (Other); Pharmacosmos A/S (Industry)
Responsible Party: Sponsor-Investigator, Michael Kremke, Principal Investigator, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICS-01
Record Dates: First submitted 2020-09-17; First posted 2020-10-29 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Anemia Postoperative
Keywords: Anemia; Iron deficiency; Transfusion; Postoperative period; Rehabilitation
MeSH Terms: conditions — Anemia; Iron Deficiencies | interventions — ferric derisomaltose; iron isomaltoside 1000; ferrous sulfate; Saline Solution

STUDY DESIGN:
Masking Description: The study is primarily open label. It includes, however, a short period (from the 1. to the 4. postoperative day) of participant, care provider and investigator masking. The aim is to reduce differences in transfusion practices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous iron group (Experimental): Single-dose intravenous infusion of 20 mg/kg body weight ferric derisomaltose/iron isomaltoside 1000 (MonoFer®)
  Interventions: Drug: Ferric Derisomaltose
- Oral iron group (Active Comparator): Oral therapy with 100 mg oral ferrous sulfate twice daily
  Interventions: Drug: Ferrous sulfate; Drug: normal saline

INTERVENTIONS:
Drug: Ferric Derisomaltose — Single-dose intravenous infusion, 20 mg/kg body weight, postoperative day 1
  Other Names: MonoFer, iron isomaltoside 1000
  Arms: Intravenous iron group
Drug: Ferrous sulfate — Oral therapy, 100 mg twice daily, from postoperative day 4 until 4-week follow-up
  Other Names: Ferro Duretter
  Arms: Oral iron group
Drug: normal saline — Single-dose infusion (placebo), postoperative day 1
  Other Names: 0.9% natriumchloride
  Arms: Oral iron group

SUMMARY:
BACKGROUND Anemia and iron deficiency are highly prevalent in cardiac surgery patients. Both conditions may adversely affect postoperative rehabilitation.

At hospital discharge, anemia is almost invariably present due to perioperative blood loss and frequent blood sampling. Two previous analyses demonstrated a prevalence of anemia early after coronary artery bypass grafting (CABG) of 94% and 98%, respectively. Almost half of CABG patients had persistent anemia two months after surgery. Postoperative anemia may result in debilitating symptoms, like dyspnoea, fatigue and poor exercise tolerance, and is associated with an increased likelihood of cardiovascular events and death after cardiac surgery.

Mild to moderate anemia is commonly corrected with oral iron supplements. Oral iron is however poorly absorbed in patients with chronic diseases, and about 40% of patients suffer from debilitating gastrointestinal side-effects. As iron stores are frequently reduced or depleted after cardiac surgery, treatment with oral iron supplements may take several months.

In patients with chronic heart failure (CHF), iron deficiency is associated with reduced exercise capacity, quality of life and survival even in the absence of anemia. Several large randomised trials demonstrated that treatment with intravenous iron improved clinical symptoms, exercise capacity and quality of life of CHF patients.

RATIONALE It is desirable to replenish body iron stores rapidly after cardiac surgery with the aim to effectively correct anemia, optimize exercise tolerance and improve patient wellbeing.

Modern intravenous iron formulations permit fast replenishment of body iron stores and have emerged as potential alternatives to oral iron. These formulations are well-tolerated and have become an established therapeutic option in anemic patients with reduced intestinal iron absorption. Several studies have demonstrated the efficacy of intravenous iron for the treatment of anemia following major non-cardiac surgery.

Data regarding the efficacy of intravenous iron in cardiac surgery, however, are conflicting.

HYPOTHESIS Single-dose intravenous iron therapy with ferric derisomaltose/iron isomaltoside is superior to oral iron supplementation for the correction of anemia following cardiac surgery. Moreover, single-dose intravenous iron therapy with ferric derisomaltose/iron isomaltoside results in a greater postoperative exercise capacity, an improved quality of life and less fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older undergoing first-time, non-emergent cardiac surgery with cardiopulmonary bypass. Eligible procedures are A: isolated CABG surgery (+/- arrhythmia surgery), B: isolated cardiac valve surgery (+/- arrhythmia surgery), C: a combination of CABG and cardiac valve surgery (+/- arrhythmia surgery)
* Moderate anaemia on the first postoperative day. According to World Health Organization-criteria defined as a haemoglobin concentration of equal to or greater than 5.0 mmol/l (8 g/dl) and less than 6.8 mmol/l (11 g/dl).

Exclusion Criteria:

* Known hypersensitivity to any iron formulation
* Multiple drug allergies or history of previous anaphylaxis
* Severe asthma, eczema or another atopic allergy
* Rheumatoid arthritis or systemic lupus erythematosus
* History of iron overload or disturbances in iron utilisation (e.g. haemochromatosis, hemosiderosis)
* History of liver disease (e.g. cirrhosis)
* Severe active infection or inflammation (e.g. endocarditis)
* Porphyria cutanea tarda
* Treatment with intravenous iron within 4 weeks prior to surgery.
* Untreated vitamin B12 or folate deficiency.
* Anticipated inability to perform a six-minute walk test.
* Women of childbearing potential, pregnant and nursing women.
* Anticipated postoperative length of stay in the intensive care unit (ICU) > 48 hours.
* Patients incapable of giving consent personally.
* Significantly increased risk of non-adherence or loss to follow-up.
* Active participation in another interventional trial with potential impact on postoperative anaemia or exercise capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
The proportion of participants who are neither anemic nor have received allogeneic red blood cells since randomisation | 4-week follow-up
  Unit: percentage; anemia according to WHO criteria defined as hemoglobin < 12 g/dl in women and < 13 g/dl in men.

SECONDARY OUTCOMES:
Mean change in hemoglobin level | From baseline to 4-week follow-up
  Unit: g/dl
Proportion of participants with a haemoglobin increase ≥ 1.3 mmol/l (≥ 2 g/dL) | From baseline to 4-week follow-up
  Unit: %
Mean haemoglobin level | 4-week follow-up
  Unit: g/dl
Mean reticulocyte count | 4-week follow-up
  Unit: 10^9/l
Mean plasma iron | 4-week follow-up
  μmol/l
Mean plasma ferritin | 4-week follow-up
  µg/l
Mean transferrin saturation | 4-week follow-up
  Unit: %
Mean change in haemoglobin level | From the day before surgery to 4-week follow-up
  Unit: g/dl
Mean change in reticulocyte count | From the day before surgery to 4-week follow-up
  Unit: 10^9/l
Mean change in plasma iron | From the day before surgery to 4-week follow-up
  μmol/l
Mean change in plasma ferritin | From the day before surgery to 4-week follow-up
  µg/l
Mean change in transferrin saturation | From the day before surgery to 4-week follow-up
  Unit: %
Proportion of participants transfused with allogeneic red blood cells | From the time of randomisation to 4-week follow-up
  Units: %
Six-minute walk distance | 4-week follow-up
  Units: meter
Health-related quality of life | 4-week follow-up
  Health-related quality of life is assessed with the standardized European Quality of Life (EuroQol) Group five dimensions questionnaire (EQ-5D). The outcome of interest is the visual analogue scale (EQ VAS). The 5-level EQ-5D (EQ-5D-5L) consists of a descriptive system and the EQ VAS. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the best endpoint is "100" and the worst "0".
Fatique | 4-week follow-up
  Fatigue is assessed using the validated Multidimensional Fatigue Inventory (MFI-20). The outcome of interest is physical fatigue. The MFI-20 consists of 20 items for the assessment of fatigue in five different dimensions: general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue. Each dimension contains four items for which participants have to indicate on a five-point scale how the particular statement suited their experience. An equal number of items are worded in a positive and a negative way to counteract for response tendencies. A score of four indicates no presence of fatigue, while a score of 20 indicates the highest level of fatigue.
New York Heart Association (NYHA) functional class | 4-week follow-up
  Assessing symptoms (i.e. angina and dyspnea) and the resulting limitations during ordinary physical activity. Class I-IV. I=no symptoms, higher classes are associated with more severe symptoms and limitations. IV=severe symptoms and limitations. The outcome of interest is the proportion of participants with a NYHA functional class of I.

OTHER OUTCOMES:
Gastrointestinal symptoms | 4-week follow-up
  Participants are asked to report the gastrointestinal symptoms the week prior to follow-up.
  We developed a simple scoring system with the five dimensions nausea, constipation, diarrhea, abdominal pain and bloating. Participants are asked to rate the presence and severity of each symptom on a scale from 0 to 3, where 0 indicates 'symptom has not been present', 1 'the symptom was present and resulted in mild discomfort', 2 '...
  moderate discomfort' and 3 '... severe discomfort'. A final score is calculated by adding each item, "15" is the worst, "0" the best outcome.
Treatment adherence to oral iron therapy | 4-week follow-up
  Units: %. Treatment adherence is measured as the proportion of oral iron tablets that the participant actually has taken in relation to the total number of tablets prescribed.
Cost-effectiveness analysis | 4-week follow-up
  Patient-specific data for resource usage are collected. Hospital resources are recorded for each individual patient from the time of randomisation until follow-up visit four weeks postoperatively:
  * study drug costs
  * units of allogeneic red blood cell transfused
  * length of hospital stay (in days)
  * length of stay in the intensive care unit (in days)
  * readmission to hospital (in days)
  * visits to outpatient clinic Costs associated with health care utilization are calculated by multiplying volumes of resources used by unit costs of that item.
Quality of Recovery Score (QoR9-questionnaire) | 4-week follow-up
  Quality of recovery (QoR) is assessed with the QoR-9 questionnaire. The QoR-9 is a patient rated score developed and validated to measure the quality of recovery after surgery and anaesthesia. This nine item instrument can be completed by patients in less than two minutes, has a maximum score of 18 and a minimum score of 0. Lesser scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kremke, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hogan M, Klein AA, Richards T. The impact of anaemia and intravenous iron replacement therapy on outcomes in cardiac surgery. Eur J Cardiothorac Surg. 2015 Feb;47(2):218-26. doi: 10.1093/ejcts/ezu200. Epub 2014 May 13. PMID 24824650
- [Background] Tramarin R, Pistuddi V, Maresca L, Pavesi M, Castelvecchio S, Menicanti L, de Vincentiis C, Ranucci M; Surgical and Clinical Outcome Research (SCORE) Group. Patterns and determinants of functional and absolute iron deficiency in patients undergoing cardiac rehabilitation following heart surgery. Eur J Prev Cardiol. 2017 May;24(8):799-807. doi: 10.1177/2047487317689975. Epub 2017 Jan 24. PMID 28117617
- [Background] Westenbrink BD, Kleijn L, de Boer RA, Tijssen JG, Warnica WJ, Baillot R, Rouleau JL, van Gilst WH; IMAGINE Investigators. Sustained postoperative anaemia is associated with an impaired outcome after coronary artery bypass graft surgery: insights from the IMAGINE trial. Heart. 2011 Oct;97(19):1590-6. doi: 10.1136/heartjnl-2011-300118. Epub 2011 Jul 13. PMID 21757458
- [Background] Ranucci M, La Rovere MT, Castelvecchio S, Maestri R, Menicanti L, Frigiola A, D'Armini AM, Goggi C, Tramarin R, Febo O. Postoperative anemia and exercise tolerance after cardiac operations in patients without transfusion: what hemoglobin level is acceptable? Ann Thorac Surg. 2011 Jul;92(1):25-31. doi: 10.1016/j.athoracsur.2011.02.058. Epub 2011 May 18. PMID 21592458
- [Background] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Brown JR, Despotis GJ, Hammon JW, Reece TB, Saha SP, Song HK, Clough ER; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Shore-Lesserson LJ, Goodnough LT, Mazer CD, Shander A, Stafford-Smith M, Waters J; International Consortium for Evidence Based Perfusion; Baker RA, Dickinson TA, FitzGerald DJ, Likosky DS, Shann KG. 2011 update to the Society of Thoracic Surgeons and the Society of Cardiovascular Anesthesiologists blood conservation clinical practice guidelines. Ann Thorac Surg. 2011 Mar;91(3):944-82. doi: 10.1016/j.athoracsur.2010.11.078. PMID 21353044
- [Background] Task Force on Patient Blood Management for Adult Cardiac Surgery of the European Association for Cardio-Thoracic Surgery (EACTS) and the European Association of Cardiothoracic Anaesthesiology (EACTA); Boer C, Meesters MI, Milojevic M, Benedetto U, Bolliger D, von Heymann C, Jeppsson A, Koster A, Osnabrugge RL, Ranucci M, Ravn HB, Vonk ABA, Wahba A, Pagano D. 2017 EACTS/EACTA Guidelines on patient blood management for adult cardiac surgery. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):88-120. doi: 10.1053/j.jvca.2017.06.026. Epub 2017 Sep 30. No abstract available. PMID 29029990
- [Background] Mazer CD, Whitlock RP, Fergusson DA, Belley-Cote E, Connolly K, Khanykin B, Gregory AJ, de Medicis E, Carrier FM, McGuinness S, Young PJ, Byrne K, Villar JC, Royse A, Grocott HP, Seeberger MD, Mehta C, Lellouche F, Hare GMT, Painter TW, Fremes S, Syed S, Bagshaw SM, Hwang NC, Royse C, Hall J, Dai D, Mistry N, Thorpe K, Verma S, Juni P, Shehata N; TRICS Investigators and Perioperative Anesthesia Clinical Trials Group. Six-Month Outcomes after Restrictive or Liberal Transfusion for Cardiac Surgery. N Engl J Med. 2018 Sep 27;379(13):1224-1233. doi: 10.1056/NEJMoa1808561. Epub 2018 Aug 26. PMID 30146969
- [Background] Tolkien Z, Stecher L, Mander AP, Pereira DI, Powell JJ. Ferrous sulfate supplementation causes significant gastrointestinal side-effects in adults: a systematic review and meta-analysis. PLoS One. 2015 Feb 20;10(2):e0117383. doi: 10.1371/journal.pone.0117383. eCollection 2015. PMID 25700159
- [Background] Piednoir P, Allou N, Driss F, Longrois D, Philip I, Beaumont C, Montravers P, Lasocki S. Preoperative iron deficiency increases transfusion requirements and fatigue in cardiac surgery patients: a prospective observational study. Eur J Anaesthesiol. 2011 Nov;28(11):796-801. doi: 10.1097/EJA.0b013e32834ad97b. PMID 21885979
- [Background] Camaschella C. Iron-deficiency anemia. N Engl J Med. 2015 May 7;372(19):1832-43. doi: 10.1056/NEJMra1401038. No abstract available. PMID 25946282
- [Background] Jankowska EA, Malyszko J, Ardehali H, Koc-Zorawska E, Banasiak W, von Haehling S, Macdougall IC, Weiss G, McMurray JJ, Anker SD, Gheorghiade M, Ponikowski P. Iron status in patients with chronic heart failure. Eur Heart J. 2013 Mar;34(11):827-34. doi: 10.1093/eurheartj/ehs377. Epub 2012 Nov 23. PMID 23178646
- [Background] von Haehling S, Ebner N, Evertz R, Ponikowski P, Anker SD. Iron Deficiency in Heart Failure: An Overview. JACC Heart Fail. 2019 Jan;7(1):36-46. doi: 10.1016/j.jchf.2018.07.015. Epub 2018 Dec 12. PMID 30553903
- [Background] Enjuanes C, Klip IT, Bruguera J, Cladellas M, Ponikowski P, Banasiak W, van Veldhuisen DJ, van der Meer P, Jankowska EA, Comin-Colet J. Iron deficiency and health-related quality of life in chronic heart failure: results from a multicenter European study. Int J Cardiol. 2014 Jun 15;174(2):268-75. doi: 10.1016/j.ijcard.2014.03.169. Epub 2014 Apr 3. PMID 24768464
- [Background] Anker SD, Comin Colet J, Filippatos G, Willenheimer R, Dickstein K, Drexler H, Luscher TF, Bart B, Banasiak W, Niegowska J, Kirwan BA, Mori C, von Eisenhart Rothe B, Pocock SJ, Poole-Wilson PA, Ponikowski P; FAIR-HF Trial Investigators. Ferric carboxymaltose in patients with heart failure and iron deficiency. N Engl J Med. 2009 Dec 17;361(25):2436-48. doi: 10.1056/NEJMoa0908355. Epub 2009 Nov 17. PMID 19920054
- [Background] Ponikowski P, van Veldhuisen DJ, Comin-Colet J, Ertl G, Komajda M, Mareev V, McDonagh T, Parkhomenko A, Tavazzi L, Levesque V, Mori C, Roubert B, Filippatos G, Ruschitzka F, Anker SD; CONFIRM-HF Investigators. Beneficial effects of long-term intravenous iron therapy with ferric carboxymaltose in patients with symptomatic heart failure and iron deficiencydagger. Eur Heart J. 2015 Mar 14;36(11):657-68. doi: 10.1093/eurheartj/ehu385. Epub 2014 Aug 31. PMID 25176939
- [Background] Okonko DO, Grzeslo A, Witkowski T, Mandal AK, Slater RM, Roughton M, Foldes G, Thum T, Majda J, Banasiak W, Missouris CG, Poole-Wilson PA, Anker SD, Ponikowski P. Effect of intravenous iron sucrose on exercise tolerance in anemic and nonanemic patients with symptomatic chronic heart failure and iron deficiency FERRIC-HF: a randomized, controlled, observer-blinded trial. J Am Coll Cardiol. 2008 Jan 15;51(2):103-12. doi: 10.1016/j.jacc.2007.09.036. PMID 18191732
- [Background] van Veldhuisen DJ, Ponikowski P, van der Meer P, Metra M, Bohm M, Doletsky A, Voors AA, Macdougall IC, Anker SD, Roubert B, Zakin L, Cohen-Solal A; EFFECT-HF Investigators. Effect of Ferric Carboxymaltose on Exercise Capacity in Patients With Chronic Heart Failure and Iron Deficiency. Circulation. 2017 Oct 10;136(15):1374-1383. doi: 10.1161/CIRCULATIONAHA.117.027497. Epub 2017 Jul 12. PMID 28701470
- [Derived] Modrau IS, Kremke M. Post-operative iron in cardiac surgery trial - a protocol for a randomised controlled trial. Dan Med J. 2022 Jun 24;69(7):A12210952. PMID 35781129